CLINICAL TRIAL: NCT01984996
Title: Freedom Inguinal Hernia Repair System Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Company was dissolved.
Sponsor: Insightra Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P0069
Record Dates: First submitted 2013-11-04; First posted 2013-11-15 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-01

CONDITIONS: Primary Inguinal Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Freedom ProFlor Inguinal Hernia Implant (Experimental)
  Interventions: Device: Freedom ProFlor Inguinal Hernia Implant

INTERVENTIONS:
Device: Freedom ProFlor Inguinal Hernia Implant

SUMMARY:
The primary objective of this study is to evaluate patient quality-of-life (QOL) after inguinal hernia repair. "Carolinas Comfort Scale" (CCS) assessments will be held at regular intervals.

The secondary objective of the study is to follow short-term and long-term study-related complications/adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo routine inguinal hernia repair
* Competent to give consent
* Clinically relevant inguinal hernia (classification: NYHUS I, II, IIIa)
* Defect size at operation is between 5mm and 35mm
* Diagnosed with unilateral, direct, indirect or mixed inguinal hernia
* Primary hernia at the operative site
* Male or female
* Life expectancy of at least 12 months
* At least 18 years of age

Exclusion Criteria:

* Signs of obvious local or systemic infection
* Any previous surgery on the hernia operative site
* Hernia is not in the inguinal area
* Hernia is not identified as indirect or direct
* Femoral hernias
* Known collagen disorder
* Presenting with unstable angina or NYHA class of IV
* Known Pregnancy
* Active drug user
* Recurrence of a repair by any method
* Patients with giant inguinoscrotal hernia or abdominal wall defect >35 mm in diameter - e.g. large direct or combined inguinal hernia type Nyhus IIIb / EHS P L/M 1/2/3
* Immunosuppression, prednisone>15 mg/day, active chemotherapy
* End stage renal disease
* Abdominal ascites
* Skin infection in area of surgical field
* BMI >35
* Peritoneum cannot be closed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Measure changes from baseline in Carolina Comfort Scale (CCS) scores at specified time intervals | 1 week, 3, 6, 9, 12, 18, 24, and 36 months.
  Measure quality of life for patients undergoing inguinal hernia repair.

SECONDARY OUTCOMES:
Evaluate the 14-day pain and medication log | 14 days
  Patient will record pain score and medications for 14 consecutive days.

OTHER OUTCOMES:
Study-related complications/adverse events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Karl LeBlanc, M.D., M.B.A., F.A.C.S., Principal Investigator — Our Lady of the Lake Hospital
Locations (8):
- United States (4):
  - Metabolic Clinic and Research Center, Los Angeles, California
  - Witham Health Services, Lebanon, Indiana
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - New Hannover Regional Medical Center, Wilmington, North Carolina
- Herz Jesu Krankenhaus GmbH, Vienna, Austria
- Italy (3):
  - Istituto Clinico Sant'Ambrogio, Milan
  - Azienda Policlinico Umberto I, Roma
  - Policlinico Tor Vergata, Roma